CLINICAL TRIAL: NCT03884101
Title: A Phase 3 Randomized, Open-Label, Study of Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) Versus Chemotherapy for First-line Treatment of Advanced or Recurrent Endometrial Carcinoma (LEAP-001)
Brief Title: Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) Versus Chemotherapy for Endometrial Carcinoma (ENGOT-en9 / MK-7902-001)
Acronym: LEAP-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-001; MK-7902-001 (Other: MSD); ENGOT-en9 (Other: European Network for Gynaecological Oncological Trial groups); 194710 (Registry Identifier: JAPIC-CTI); 2023-505614-17-00 (Registry Identifier: EU CT); U1111-1292-1245 (Registry Identifier: UTN); 2018-003009-24 (EudraCT Number)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib; pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib + Pembrolizumab (Experimental): Participants receive lenvatinib daily and pembrolizumab once at the start of each 3-week treatment cycle.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- Paclitaxel + Carboplatin (Active Comparator): Participants receive paclitaxel and carboplatin once at the start of each 3-week treatment cycle.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 4 mg or 10 mg capsules at a total daily dose of 20 mg taken by mouth once per day.
  Other Names: E7080, MK-7902, LENVIMA®
  Arms: Lenvatinib + Pembrolizumab
Biological: Pembrolizumab — Pembrolizumab 200 mg intravenous (IV) infusion given on Day 1 of each cycle.
  Other Names: MK-3475, KEYTRUDA®
  Arms: Lenvatinib + Pembrolizumab
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 IV infusion given on Day 1 of each cycle.
  Other Names: TAXOL®, ONXAL®
  Arms: Paclitaxel + Carboplatin
Drug: Carboplatin — Carboplatin 10 mg/mL IV infusion at a total dose of are-under-the-curve (AUC) 6 (per Calvert's formula) given on Day 1 of each cycle.
  Other Names: PARAPLATIN®
  Arms: Paclitaxel + Carboplatin

SUMMARY:
The purpose of this study is to compare the efficacy of pembrolizumab + lenvatinib to chemotherapy in female participants with Stage III, IV, or recurrent endometrial carcinoma. It is hypothesized that the combination of pembrolizumab + lenvatinib will be superior to chemotherapy for progression-free survival (PFS) per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR). It is also hypothesized that the combination of pembrolizumab + lenvatinib will be superior to chemotherapy for overall survival (OS).

As of Amendment 7 eligible participants on study completion will be able to transition to an extension study, if available, in which they can continue to receive pembrolizumab monotherapy, lenvatinib monotherapy, or a combination of both pembrolizumab and lenvatinib as received in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Has Stage III, Stage IV, or recurrent, histologically-confirmed endometrial carcinoma with disease that is either measurable or nonmeasurable but radiographically apparent, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR) (note: may have received prior chemotherapy only if administered concurrently with radiation; may have received prior radiation without concurrent chemotherapy; may have received prior hormonal therapy for treatment of endometrial carcinoma, provided that it was discontinued ≥1 week prior to randomization; and may have received 1 prior line of systemic platinum-based adjuvant and/or neoadjuvant chemotherapy)
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion that was not previously irradiated, for determination of mismatch repair (MMR) status
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 7 days prior to the first dose of study intervention
* Is not pregnant or breastfeeding, and is either not a woman of childbearing potential (WOCBP) or is a WOCBP who agrees to use contraception during the study and for ≥120 days after pembrolizumab, ≥30 days after lenvatinib, or ≥180 days after (chemotherapy) [if a WOCBP, a pregnancy test will be required within 24 hours of first dose of study drug]
* Has adequately controlled blood pressure within 7 days prior to randomization
* Has adequate organ function based on assessment within 7 days prior to the first dose of study intervention

Exclusion Criteria:

* Has carcinosarcoma (malignant mixed Műllerian tumor), endometrial leiomyosarcoma or other high grade sarcomas, or endometrial stromal sarcomas
* Has a central nervous system (CNS) metastasis, unless local therapy (e.g., whole brain radiation therapy, surgery, or radiosurgery) has been completed and have discontinued use of corticosteroids for this indication for ≥4 weeks prior to starting study medication (major surgery within 3 weeks of the first dose of study drug will be exclusionary)
* Has a known additional malignancy (other than endometrial carcinoma) that is progressing or has required active treatment in the last 3 years
* Has gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
* Has a pre-existing Grade ≥3 gastrointestinal or nongastrointestinal fistula
* Has radiographic evidence of major blood vessel invasion/infiltration
* Has active hemoptysis (bright red blood at ≥0.5 teaspoon) within 3 weeks prior to the first dose of study intervention or tumor bleeding within 2 weeks prior to randomization
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction or cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has any infection requiring systemic treatment
* Has not recovered adequately from any toxicity and/or complications from major surgery prior to randomization
* Has a known history of human immunodeficiency virus (HIV) infection (HIV test is required at screening)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) [defined as HCV ribonucleic acid (RNA) is detected] (hepatitis B and C testing is required at screening only when mandated by local health authority)
* Has a history of (noninfectious) pneumonitis that required treatment with steroids, or has current pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has an active autoimmune disease (with the exception of psoriasis) that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has received prior systemic chemotherapy in any setting for the treatment of endometrial carcinoma (note: prior chemotherapy administered concurrently with radiation is permitted)
* Has received prior radiotherapy within 4 weeks prior to randomization (participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis - a 2-week washout is permitted for palliative radiation to non-CNS disease and vaginal brachytherapy)
* Has received prior hormonal therapy for the treatment of endometrial carcinoma within 1 week of randomization
* Has received prior therapy with any treatment targeting vascular endothelial growth factor (VEGF)-directed angiogenesis, an anti-programmed cell death (PD)-1, anti-PD ligand (L)1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Has known intolerance to study intervention (or any of the excipients)
* Has had an allogenic tissue/solid organ transplant
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (195):
- United States (29):
  - University of South Alabama, Mitchell Cancer Institute ( Site 0245), Mobile, Alabama
  - Arizona Oncology Associates PC- HOPE ( Site 8005), Tucson, Arizona
  - UCLA Hematology and Oncology Clinic (Westwood) ( Site 0233), Los Angeles, California
  - University of Colorado Cancer Center ( Site 0204), Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven ( Site 0202), New Haven, Connecticut
  - University of Miami Health System ( Site 0249), Miami, Florida
  - Georgia Cancer Center at Augusta University ( Site 0222), Augusta, Georgia
  - Women's Cancer Care ( Site 0208), Covington, Louisiana
  - Maine Medical Partners ( Site 0217), Scarborough, Maine
  - Minnesota Oncology Hematology, PA ( Site 8003), Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Center At Basking Ridge ( Site 0268), Basking Ridge, New Jersey
  - John Theurer Cancer Center at Hackensack University Med Ctr ( Site 0226), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 0273), Middletown, New Jersey
  - MSKCC-Bergen ( Site 0276), Montvale, New Jersey
  - Holy Name Medical Center ( Site 0235), Teaneck, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 0267), Commack, New York
  - Memorial Sloan Kettering Cancer Center - West Harrison ( Site 0274), Harrison, New York
  - The Blavatnik Family- Chelsea Medical Center at Mount Sinai ( Site 0206), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0246), New York, New York
  - University of Rochester ( Site 0238), Rochester, New York
  - Memorial Sloan Kettering Cancer Center - Nassau ( Site 0275), Uniondale, New York
  - University of North Carolina- Chapel Hill ( Site 0254), Chapel Hill, North Carolina
  - Roger Maris Cancer Center ( Site 0277), Fargo, North Dakota
  - Willamette Valley Cancer Institute and Research Center ( Site 8004), Eugene, Oregon
  - Sanford Cancer Center Oncology Clinic ( Site 0205), Sioux Falls, South Dakota
  - Parkland Health & Hospital System ( Site 0272), Dallas, Texas
  - University of Texas Southwestern Medical Center ( Site 0264), Dallas, Texas
  - Texas Oncology-The Woodlands ( Site 8000), The Woodlands, Texas
  - Legacy Salmon Creek Medical Center ( Site 0253), Vancouver, Washington
- Argentina (6):
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 2607), Caba, Buenos Aires
  - Hospital Italiano de La Plata ( Site 2601), La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 2606), Mar del Plata, Buenos Aires
  - Hospital Aleman ( Site 2600), Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 2603), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 2605), La Rioja
- Australia (8):
  - Chris OBrien Lifehouse ( Site 1605), Camperdown, New South Wales
  - Prince of Wales Hospital [Australia] ( Site 1603), Randwick, New South Wales
  - Royal North Shore Hospital ( Site 1600), St Leonards, New South Wales
  - The Crown Princess Mary Cancer Centre - Westmead Hospital ( Site 1602), Westmead, New South Wales
  - Mater Misericordiae Ltd ( Site 1608), South Brisbane, Queensland
  - Monash Health ( Site 1606), Clayton, Victoria
  - Epworth Freemasons Hospital ( Site 1609), Melbourne, Victoria
  - Sir Charles Gairdner Hospital ( Site 1604), Nedlands, Western Australia
- Austria (3):
  - Universitatsklinik fuer Frauenheilkunde und Geburtshilfe ( Site 3301), Graz, Styria
  - Medizinische Universitat Innsbruck ( Site 3302), Innsbruck, Tyrol
  - Medizinische Universitat Wien ( Site 3300), Vienna, Vienna
- Belgium (5):
  - UZA University Hospital Antwerp ( Site 3204), Edegem, Antwerpen
  - UZ Leuven ( Site 3200), Leuven, Antwerpen
  - Cliniques Universitaires Saint-Luc ( Site 3203), Brussels, Bruxelles-Capitale, Region de
  - AZ Maria Middelares Gent ( Site 3202), Ghent, Oost-Vlaanderen
  - AZ Delta ( Site 3206), Roeselare, West-Vlaanderen
- Brazil (10):
  - Instituto do Cancer do Ceara ( Site 2703), Fortaleza, Ceará
  - Hospital Araujo Jorge Associacao de Combate ao Cancer de Goias ( Site 2702), Goiânia, Goiás
  - Faculdade de Medicina da Universidade Federal de Minas Gerais ( Site 2708), Belo Horizonte, Minas Gerais
  - Hospital de Caridade de Ijui ( Site 2712), Ijuí, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 2701), Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose de Rio Preto ( Site 2704), São José do Rio Preto, São Paulo
  - Instituto Nacional do Cancer II ( Site 2707), Rio de Janeiro
  - Clinica de Pesquisas e Ctro de Estudos Onc. Ginecol. e Mamaria Ltda ( Site 2706), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 2713), São Paulo
  - A.C. Camargo Cancer Center ( Site 2705), São Paulo
- Canada (12):
  - Cross Cancer Institute ( Site 0408), Edmonton, Alberta
  - BC Cancer-Kelowna - Sindi Ahluwalia Hawkins Centre ( Site 0402), Kelowna, British Columbia
  - BC Cancer-Vancouver Center ( Site 0412), Vancouver, British Columbia
  - Juravinski Cancer Centre ( Site 0406), Hamilton, Ontario
  - Kingston Health Sciences Centre ( Site 0401), Kingston, Ontario
  - The Credit Valley Hospital ( Site 0403), Mississauga, Ontario
  - Sunnybrook Research Institute ( Site 0410), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0409), Toronto, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0414), Montreal, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0411), Montreal, Quebec
  - McGill University Health Centre ( Site 0404), Montreal, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0417), Sherbrooke, Quebec
- China (16):
  - Anhui Provincial Cancer Hospital ( Site 2509), Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital Capital Medical University ( Site 2505), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 2501), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 2504), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 2513), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital.Sun Yat-sen University ( Site 2507), Guangzhou, Guangdong
  - Guang Xi Tumour Hospital, Department of Chemotherapy ( Site 2517), Nanning, Guangxi
  - Hubei Cancer Hospital ( Site 2510), Wuhan, Hubei
  - Xiangya Hospital Central-South University ( Site 2512), Changsha, Hunan
  - Nanjing Maternity and Child Health Care Hospital ( Site 2508), Nanjing, Jiangsu
  - The first affiliated Hospital of Xi an Jiaotong University ( Site 2502), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center ( Site 2500), Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hosp. Fudan University ( Site 2503), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University ( Site 2515), Ürümqi, Xinjiang
  - Women s Hospital School of Medicine Zhejiang University ( Site 2511), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2506), Hangzhou, Zhejiang
- Germany (7):
  - Universitaetsmedizin Mannheim. Klinik fuer Kinder und Jugendmedizin ( Site 0622), Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Muenster ( Site 0615), Münster, Baden-Wurttemberg
  - Caritas-Krankenhaus St. Josef Regensburg ( Site 0613), Regensburg, Bavaria
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden ( Site 0623), Wiesbaden, Hesse
  - Universitaetsklinikum Essen ( Site 0616), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Jena ( Site 0612), Jena, Thuringia
  - Charite Universitaetsmedizin Berlin ( Site 0609), Berlin
- Ireland (2):
  - Cork University Hospital ( Site 1400), Cork
  - St James Hospital ( Site 1401), Dublin
- Israel (4):
  - Meir Medical Center ( Site 0702), Kfar Saba, Central District
  - Edith Wolfson Medical Center ( Site 0703), Holon, Tell Abib
  - Rambam Medical Center ( Site 0700), Haifa
  - Chaim Sheba Medical Center ( Site 0707), Ramat Gan
- Italy (9):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 0800), Meldola, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli ( Site 0805), Rome, Roma
  - Ospedale dell Angelo ( Site 0810), Mestre, Venezia
  - Medical Oncology Ospedale San Donato ( Site 0812), Arezzo
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 0801), Bari
  - Ospedale Policlinico S. Orsola-Malpighi ( Site 0803), Bologna
  - Ospedale Antonio Perrino ( Site 0806), Brindisi
  - Azienda Ospedaliera per l Emergenza Cannizzaro ( Site 0807), Catania
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0808), Napoli
- Japan (18):
  - Ehime University Hospital ( Site 2413), Tōon, Ehime
  - Kurume University Hospital ( Site 2403), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 2404), Ōta, Gunma
  - National Hospital Organization Hokkaido Cancer Center ( Site 2408), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 2414), Akashi, Hyōgo
  - Nippon Medical School Musashi Kosugi Hospital ( Site 2417), Kawasaki, Kanagawa
  - St. Marianna University School of Medicine Hospital ( Site 2416), Kawasaki, Kanagawa
  - University of the Ryukyus Hospital ( Site 2412), Nakagami-gun, Okinawa
  - Saitama Medical University International Medical Center ( Site 2410), Hidaka, Saitama
  - Saitama Cancer Center ( Site 2406), Kitaadachi-gun, Saitama
  - National Defense Medical College Hospital ( Site 2418), Tokorozawa, Saitama
  - Kyorin University Hospital ( Site 2402), Mitaka, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 2405), Fukuoka
  - Niigata Cancer Center Hospital ( Site 2415), Niigata
  - Osaka International Cancer Institute ( Site 2409), Osaka
  - The Cancer Institute Hospital of JFCR ( Site 2401), Tokyo
  - Showa University Hospital ( Site 2419), Tokyo
  - Keio University Hospital ( Site 2411), Tokyo
- Mexico (6):
  - Hospital San Lucas Cardiologica del Sureste ( Site 3103), Tuxtla Gutiérrez, Chiapas
  - I CAN Oncology SA de SV ( Site 3102), Monterrey, Nuevo León
  - Centro Estatal de Cancerologia de Chihuahua ( Site 3101), Chihuahua City
  - Centro de Investigacion Clinica Gramel ( Site 3107), Mexico City
  - Centro Oncologico Internacional. SEDNA ( Site 3106), Mexico City
  - Consultorio Dentro de la Torre Medica Dalinde Oncologia Medica ( Site 3108), Mexico City
- Poland (8):
  - Wielkopolskie Centrum Onkologii im.M.Sklodowskiej-Curie ( Site 1004), Poznan, Greater Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 1019), Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie ( Site 1008), Lublin, Lower Silesian Voivodeship
  - Szpital Kliniczny im Ks Anny Mazowieckiej ( Site 1011), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 1009), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1005), Bialystok, Podlaskie Voivodeship
  - Centrum Onkologii Instytut im. MSC Oddział w Gliwicach ( Site 1017), Gliwice, Silesian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki ( Site 1020), Lodz, Łódź Voivodeship
- Russia (11):
  - Krasnoyarsk Regional Clinical oncology dispensary ( Site 1118), Krasnoyarsk, Krasnoyarsk Krai
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 1100), Moscow, Moscow
  - FSBI-FRCC of Special Types Med. Care and Technologies FMBA of Russia ( Site 1102), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 1101), Moscow, Moscow
  - Samara Regional Clinical Oncology Center ( Site 1117), Samara, Samara Oblast
  - St.Petersburg Clinical Hospital RAS ( Site 1124), Saint Petersburg, Sankt-Peterburg
  - Railway Hospital of OJSC ( Site 1122), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 1103), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City Clinical Oncological Dispensary ( Site 1104), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1108), Kazan', Tatarstan, Respublika
  - Siberian State Medical University ( Site 1121), Tomsk, Tomsk Oblast
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 1802), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 1801), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1804), Seoul
  - Asan Medical Center ( Site 1800), Seoul
  - Samsung Medical Center ( Site 1803), Seoul
- Spain (8):
  - Institut Catala d Oncologia Badalona ( Site 1201), Badalona, Barcelona
  - Complejo Hospitalario Universitario A Coruna. CHUAC ( Site 1202), A Coruña, La Coruna
  - Instituto Valenciano de Oncologia - IVO ( Site 1205), Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Valencia ( Site 1203), Valencia, Valenciana, Comunitat
  - Parc de Salut Mar ( Site 1200), Barcelona
  - Hospital Universitario Reina Sofia ( Site 1207), Córdoba
  - Hospital Clinico San Carlos ( Site 1209), Madrid
  - Hospital Materno Infantil [Malaga, Spain] ( Site 1208), Málaga
- Taiwan (5):
  - China Medical University Hospital ( Site 1903), Taichung
  - Taichung Veterans General Hospital ( Site 1902), Taichung
  - National Taiwan University Hospital ( Site 1904), Taipei
  - Taipei Veterans General Hospital ( Site 1900), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 1901), Taoyuan District
- Turkey (Türkiye) (6):
  - Baskent Universitesi Adana Uygulama ve Arastirma Hastanesi ( Site 1303), Adana
  - Cukurova Uni. Tip Fakultesi ( Site 1302), Adana
  - Gazi Universitesi Tip Fakultesi ( Site 1308), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 1300), Ankara
  - Akdeniz Universitesi Tıp Fakultesi ( Site 1301), Antalya
  - Uludag Universitesi Tip Fakultesi ( Site 1307), Bursa
- Ukraine (11):
  - Clinical oncology dispensary of Dnipro ( Site 1512), Dnipro, Dnipropetrovsk Oblast
  - City Clinical Hosp.4 of DCC ( Site 1501), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 1503), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 1511), Kharkiv, Kharkivs’ka Oblast’
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1509), Kharkiv, Kharkivs’ka Oblast’
  - Khmelnitskiy Regional Onkology Dispensary ( Site 1513), Khmelnitskiy, Khmelnytskyi Oblast
  - Medical Center Asklepion LLC ( Site 1514), Khodosovka, Kyivska Oblast
  - National Cancer Institute of the MoH of Ukraine ( Site 1510), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 1507), Kyiv, Kyivska Oblast
  - MI Odessa Regional Oncological Centre ( Site 1504), Odesa, Odesa Oblast
  - Kyiv City Clinical Oncology Centre ( Site 1505), Kyiv
- United Kingdom (6):
  - Western General Hospital ( Site 1411), Edinburgh, Edinburgh, City of
  - UCLH NHS Foundation Trust ( Site 1405), London, London, City of
  - Mount Vernon Cancer Centre ( Site 1409), Northwood, London, City of
  - Churchill Hospital ( Site 1406), Oxford, Oxfordshire
  - The James Cook University Hospital ( Site 1403), Middlesbrough
  - Northern Centre for Cancer Care ( Site 1408), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Marth C, Moore RG, Bidzinski M, Pignata S, Ayhan A, Rubio MJ, Beiner M, Hall M, Vulsteke C, Braicu EI, Sonoda K, Wu X, Frentzas S, Mattar A, Lheureux S, Chen X, Hasegawa K, Magallanes-Maciel M, Choi CH, Shalkova M, Kaen D, Wang PH, Berger R, Okpara CE, McKenzie J, Yao L, Orlowski R, Khemka V, Gilbert L, Makker V; ENGOT-en9/LEAP-001 Investigators. First-Line Lenvatinib Plus Pembrolizumab Versus Chemotherapy for Advanced Endometrial Cancer: A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2025 Mar 20;43(9):1083-1100. doi: 10.1200/JCO-24-01326. Epub 2024 Nov 26. PMID 39591551
- [Derived] Marth C, Moore RG, Bidzinski M, Salutari V, Altundag O, Rubio MJ, Levy T, Stillie A, Vulsteke C, Witteler R, Ariyoshi K, Wu X, Frentzas S, Mattar A, Slomovitz BM, Lheureux S, Chen X, Hasegawa K, Magallanes M, Choi CH, Shalkova M, Kaen DL, Cadoo K, Yao L, McKenzie J, Okpara CE, Meng R, Orlowski R, Gilbert L, Makker V. First-line lenvatinib plus pembrolizumab versus chemotherapy for advanced endometrial cancer: 1-Year follow-up after final analysis of the ENGOT-en9/LEAP-001 phase 3 trial. Int J Gynecol Cancer. 2026 Jan;36(1):102795. doi: 10.1016/j.ijgc.2025.102795. Epub 2025 Nov 11. PMID 41494216
- [Derived] Marth C, Tarnawski R, Tyulyandina A, Pignata S, Gilbert L, Kaen D, Rubio MJ, Frentzas S, Beiner M, Magallanes-Maciel M, Farrelly L, Choi CH, Berger R, Lee C, Vulsteke C, Hasegawa K, Braicu EI, Wu X, McKenzie J, Lee JJ, Makker V. Phase 3, randomized, open-label study of pembrolizumab plus lenvatinib versus chemotherapy for first-line treatment of advanced or recurrent endometrial cancer: ENGOT-en9/LEAP-001. Int J Gynecol Cancer. 2022 Jan;32(1):93-100. doi: 10.1136/ijgc-2021-003017. Epub 2021 Nov 19. PMID 34799418
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26245&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 842 total participants randomized in the MK-7902-001 global study, 66 were also randomized in the China extension study for MK-7902-001 (NCT04865289).
Pre-assignment Details: Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Lenvatinib + Pembrolizumab: Participants received lenvatinib 20 mg orally daily until disease progression or toxicity and pembrolizumab 200 mg intravenous (IV) once at the start of each 3-week treatment cycle (Q3W) for up to 35 cycles (up to ~2 years). Eligible participants who stopped initial course of pembrolizumab plus lenvatinib and achieved Stable Disease (SD) or better but progressed after discontinuation, initiated a second course of pembrolizumab 200mg IV Q3W (for up to 17 cycles [up to ~ 1 year]) with daily lenvatinib 20 mg orally, at investigator's discretion. Treatment with lenvatinib could have been stopped at any time in the first or second course due to toxicity or disease progression.
- Paclitaxel + Carboplatin: Participants received paclitaxel 175 mg/m^2 IV Q3W and carboplatin area under the curve (AUC) 6 mg/ml/min IV Q3W once at the start of each 3-week treatment cycle for up to 7 cycles. Participants continued receiving treatment beyond 7 cycles at the investigator's discretion.
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Started | 420 | 422
Treated | 420 | 411
Received a Second Course of Pembrolizumab | 17 | 0
Completed | 0 | 0
Not Completed | 420 | 422
Not completed — Death | 234 | 248
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 98 | 126
Not completed — Sponsor Decision | 79 | 32
Not completed — Withdrawal by Subject | 8 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 420 | 422 | 842
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (10.1) | 64.0 (9.1) | 63.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 420 | 422 | 842
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 67 | 131
  Not Hispanic or Latino | 347 | 343 | 690
  Unknown or Not Reported | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 114 | 102 | 216
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 14 | 24
  White | 288 | 300 | 588
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants were stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG=0 | 250 | 240 | 490
    ECOG=1 | 170 | 182 | 352
Prior Chemotherapy and/or Chemoradiation [Count of Participants; unit: Participants] — Participants were stratified by whether or not they had received prior chemotherapy and/or chemoradiation treatment; yes or no.
  Participants
    Yes | 74 | 68 | 142
    No | 346 | 354 | 700
Mismatch Repair (MMR) Status [Count of Participants; unit: Participants] — Participants were stratified by their MMR status; Mismatch Repair Proficient (pMMR) or Mismatch Repair Deficient (dMMR).
  Participants
    dMMR | 100 | 100 | 200
    pMMR | 320 | 322 | 642

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Mismatch Repair Proficient (pMMR) Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS of pMMR participants was presented.
Time Frame: Up to approximately 44 months
Population: All randomized pMMR participants were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 320 | 322
Months | 9.6 [8.2 to 11.9] | 10.2 [8.4 to 10.4]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.5550121, Log Rank; One-sided p-value based on log-rank test and stratified by ECOG performance status and prior chemotherapy and/or chemoradiation; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.83 to 1.24] — Based on Cox regression model with Efron's method for tie handling with treatment as a covariate stratified by ECOG performance status and prior chemotherapy and/or chemoradiation

2. Primary Outcome: PFS Based on RECIST 1.1 as Assessed by BICR in All Randomized Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS of all randomized participants was presented.
Time Frame: Up to approximately 44 months
Population: All randomized participants were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 422
Months | 12.5 [10.3 to 15.1] | 10.2 [8.4 to 10.4]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.1792058, Log Rank; One-sided p-value based on log-rank test and stratified by MMR status, ECOG performance status, and prior chemotherapy and/or chemoradiation; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — Based on Cox regression model with Efron's method for tie handling with treatment as a covariate stratified by MMR status, ECOG performance status, and prior chemotherapy and/or chemoradiation

3. Primary Outcome: Overall Survival (OS) in pMMR Participants
Description: OS was measured from the time of randomization up to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The OS for pMMR participants is presented.
Time Frame: Up to approximately 51 months
Population: All randomized pMMR participants were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 320 | 322
Months | 30.9 [25.4 to 37.7] | 29.4 [26.2 to 35.4]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Non-Inferiority — The null hypothesis for the non-inferiority test was that the hazard ratio was equal to 1.1; p = 0.2459875, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.5875597, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.26] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: OS in All Randomized Participants
Description: OS was measured from the time of randomization up to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The OS for all randomized participants is presented.
Time Frame: Up to approximately 51 months
Population: All randomized participants were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 422
Months | 37.7 [32.2 to 43.6] | 32.1 [27.2 to 35.7]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.21552, Log Rank; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.12] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Objective Response Rate (ORR) Based on RECIST 1.1 as Assessed by BICR in pMMR Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of pMMR participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 51 months
Population: Per protocol, all randomized pMMR participants with measurable disease at the baseline scan were analyzed according to the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 318 | 317
Percentage of Participants | 50.9 [45.3 to 56.6] | 55.2 [49.5 to 60.8]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other; p = 0.8569, Stratified Miettinen & Nurminen; One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = -4.2, 95% CI 2-sided [-11.9 to 3.5] — Based on Miettinen & Nurminen method stratified by ECOG performance status and prior chemotherapy and/or chemoradiation

6. Secondary Outcome: ORR Based on RECIST 1.1 as Assessed by BICR in All Randomized Participants
Description: ORR was defined as the percentage of participants who had a CR: Disappearance of all target lesions or a PR: At least a 30% decrease in the sum of diameters of target lesions as assessed using RECIST 1.1. The percentage of all randomized participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 51 months
Population: Per protocol, all randomized participants with measurable disease at the baseline scan were analyzed according to the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 418 | 416
Percentage of Participants | 56.0 [51.1 to 60.8] | 56.0 [51.1 to 60.8]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other; p = 0.4999, Stratified Miettinen & Nurminen; One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 0.0, 95% CI 2-sided [-6.7 to 6.7] — Based on Miettinen & Nurminen method stratified by MMR status, ECOG performance status, and prior chemotherapy and/or chemoradiation

7. Secondary Outcome: Mean Change From Baseline in the Global Health Status/Quality of Life Score of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30) in pMMR Participants
Description: The EORTC QLQ-C30 was developed to assess the quality of life of patients with cancer. It contains 30 questions (items), 24 of which aggregate into nine multi-item scales representing various aspects, or dimensions, of quality of life (QoL): one global scale, five functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea, pain), and six additional single-symptom items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Individual items are scored on a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Raw scores for each scale are standardized into a range of 0 to 100 by linear transformation; a higher score on the global and functional scales represents a higher ("better") level of functioning, and a higher score on the symptom scale represents a higher ("worse") level of symptoms.
Time Frame: Baseline and up to approximately 18 weeks
Population: All randomized pMMR participants who had at least one assessment available for EORTC QLQ-C30 and received at least one dose of the study intervention were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 318 | 310
Scores on a scale | -5.10 [-7.76 to -2.45] | -1.34 [-4.00 to 1.32]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — Based on a constrained longitudinal data analysis (cLDA) model with the patient-reported outcome (PRO) scores as the response variable with covariates for treatment by study visit interaction, and stratification factors ECOG performance status, and prior chemotherapy and/or chemoradiation; p = 0.0302, cLDA model; Difference in Least Square Means = -3.77, 95% CI 2-sided [-7.17 to -0.36]

8. Secondary Outcome: Mean Change From Baseline in the Global Health Status/Quality of Life Score of the EORTC QLQ-C30 in All Randomized Participants
Description: The EORTC QLQ-C30 was developed to assess the quality of life of patients with cancer. It contains 30 questions (items), 24 of which aggregate into nine multi-item scales representing various aspects, or dimensions, of QoL: one global scale, five functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea, pain), and six additional single-symptom items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Individual items are scored on a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Raw scores for each scale are standardized into a range of 0 to 100 by linear transformation; a higher score on the global and functional scales represents a higher ("better") level of functioning, and a higher score on the symptom scale represents a higher ("worse") level of symptoms.
Time Frame: Baseline and up to approximately 18 weeks
Population: All randomized participants who had at least one assessment available for EORTC QLQ-C30 and received at least one dose of the study intervention were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 415 | 403
Scores on a scale | -4.52 [-6.84 to -2.20] | -2.22 [-4.60 to 0.15]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors MMR status, ECOG performance status, and prior chemotherapy and/or chemoradiation; p = 0.1355, cLDA model; Difference in Least Square Means = -2.29, 95% CI 2-sided [-5.31 to 0.72]

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). Per protocol, the number of participants who experienced one or more AEs was reported for the first course lenvatinib + pembrolizumab and paclitaxel + carboplatin arms.
Time Frame: Up to approximately 68 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Lenvatinib + Pembrolizumab: Participants received lenvatinib 20 mg orally daily until disease progression or toxicity and pembrolizumab 200 mg intravenous (IV) once at the start of each 3-week treatment cycle (Q3W) for up to 35 cycles (up to ~2 years). Eligible participants who stopped initial course of pembrolizumab plus lenvatinib and achieved Stable Disease (SD) or better but progressed after discontinuation, initiated a second course of pembrolizumab 200 mg Q3W (for up to 17 cycles [up to ~ 1 year]) with daily lenvatinib 20 mg orally daily, at investigator's discretion. Treatment with lenvatinib could have been stopped at any time in the first or second course due to toxicity or disease progression.
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 411
Participants | 418 | 405

10. Secondary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE was an AE that resulted in death, was life-threatening, required or prolonged hospitalization, resulted in persistent or significant disability, was a congenital birth defect, or was another important medical event. Per protocol, the number of participants who experienced one or more SAEs was reported for the first course lenvatinib + pembrolizumab and paclitaxel + carboplatin arms.
Time Frame: Up to approximately 68 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 411
Participants | 230 | 84

11. Secondary Outcome: Number of Participants Who Experienced an Immune-Related Adverse Event (irAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Immune-related AEs (irAEs) were AEs that were considered immune-mediated or potentially immune-mediated and are well-documented for pembrolizumab. These irAEs may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. Per protocol, the number of participants who experienced one or more irAEs was reported for the first course lenvatinib + pembrolizumab and paclitaxel + carboplatin arms.
Time Frame: Up to approximately 68 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 411
Participants | 316 | 56

12. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). Per protocol, the number of participants who discontinued any study intervention (pembrolizumab and/or lenvatinib or paclitaxel and/or carboplatin) due to an AE was reported for the first course lenvatinib + pembrolizumab and paclitaxel + carboplatin arms.
Time Frame: Up to approximately 68 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 420 | 411
Participants | 203 | 80

ADVERSE EVENTS:
Time Frame: Up to approximately 68 months
Description: All-Cause Mortality (ACM) included all randomized participants. Adverse events (AEs) included all participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment were excluded as AEs. ACM & AEs were reported separately for second course treatment.
Groups:
- First Course: Lenvatinib + Pembrolizumab: Participants received lenvatinib 20 mg orally daily until disease progression or toxicity and pembrolizumab 200 mg intravenous (IV) once at the start of each 3-week treatment cycle (Q3W) for up to 35 cycles (up to ~2 years).
- Second Course: Lenvatinib + Pembrolizumab: Eligible participants who stopped initial course of pembrolizumab plus lenvatinib and achieved Stable Disease (SD) or better but progressed after discontinuation, initiated a second course of pembrolizumab 200 mg Q3W (for up to 17 cycles [up to ~ 1 year]) with daily lenvatinib 20 mg orally, at investigator's discretion. Treatment with lenvatinib could have been stopped at any time in the first or second course due to toxicity or disease progression.
Arm/Group | First Course: Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin | Second Course: Lenvatinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 233/420 | 253/422 | 3/17
Serious Adverse Events (participants affected / at risk) | 230/420 | 84/411 | 3/17
Other Adverse Events (participants affected / at risk) | 416/420 | 397/411 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Course: Lenvatinib + Pembrolizumab (N=420) | Paclitaxel + Carboplatin (N=411) | Second Course: Lenvatinib + Pembrolizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 9 (10) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 9 (10) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia malignant (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (4) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Systemic bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (12) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 3 (4) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Assisted suicide (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 5 (6) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Course: Lenvatinib + Pembrolizumab (N=420) | Paclitaxel + Carboplatin (N=411) | Second Course: Lenvatinib + Pembrolizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 95 (130) | 209 (300) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 6 (8) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 14 (45) | 53 (149) | 1 (3)
Lymphopenia (Blood and lymphatic system disorders) | 8 (14) | 14 (29) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 19 (51) | 126 (295) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (34) | 69 (132) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (7) | 7 (7) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 71 (77) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 261 (323) | 10 (11) | 3 (4)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Scintillating scotoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 22 (26) | 11 (13) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 102 (153) | 62 (76) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 12 (12) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 51 (68) | 21 (25) | 0 (0)
Constipation (Gastrointestinal disorders) | 105 (144) | 109 (144) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 214 (568) | 97 (136) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 38 (41) | 8 (9) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 25 (32) | 15 (17) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 (23) | 18 (19) | 0 (0)
Nausea (Gastrointestinal disorders) | 159 (294) | 173 (331) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 72 (104) | 20 (30) | 2 (2)
Vomiting (Gastrointestinal disorders) | 107 (222) | 68 (95) | 1 (1)
Asthenia (General disorders) | 102 (151) | 81 (145) | 1 (1)
Chills (General disorders) | 8 (9) | 7 (8) | 2 (2)
Fatigue (General disorders) | 145 (205) | 118 (142) | 1 (1)
Influenza like illness (General disorders) | 13 (16) | 3 (3) | 1 (1)
Malaise (General disorders) | 25 (37) | 27 (46) | 0 (0)
Mucosal inflammation (General disorders) | 47 (61) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 66 (84) | 22 (22) | 1 (1)
Pain (General disorders) | 23 (23) | 18 (21) | 0 (0)
Pyrexia (General disorders) | 60 (83) | 25 (28) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 39 (42) | 5 (5) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 8 (10) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 102 (192) | 54 (76) | 3 (5)
Viral abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (12) | 5 (6) | 1 (1)
Alanine aminotransferase increased (Investigations) | 117 (209) | 45 (57) | 1 (1)
Amylase decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 42 (87) | 13 (14) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 110 (196) | 30 (38) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 57 (91) | 26 (33) | 1 (4)
Blood bilirubin increased (Investigations) | 25 (48) | 2 (2) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood cholesterol increased (Investigations) | 37 (68) | 12 (12) | 1 (1)
Blood creatinine increased (Investigations) | 50 (89) | 16 (20) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 39 (65) | 11 (13) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 33 (47) | 3 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 73 (124) | 15 (21) | 0 (0)
Lymphocyte count decreased (Investigations) | 20 (45) | 28 (44) | 0 (0)
Neutrophil count decreased (Investigations) | 25 (52) | 128 (413) | 0 (0)
Platelet count decreased (Investigations) | 50 (86) | 77 (162) | 0 (0)
Weight decreased (Investigations) | 122 (141) | 25 (26) | 1 (1)
White blood cell count decreased (Investigations) | 23 (41) | 105 (303) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 144 (206) | 82 (114) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 18 (21) | 13 (15) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 31 (40) | 13 (18) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 42 (89) | 29 (33) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 43 (94) | 11 (13) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 38 (59) | 10 (15) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 29 (40) | 13 (19) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 67 (150) | 29 (46) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 62 (112) | 68 (87) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 40 (58) | 15 (17) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 132 (192) | 97 (197) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 78 (94) | 30 (35) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 23 (42) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 24 (30) | 10 (12) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 68 (92) | 75 (122) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 63 (97) | 53 (71) | 1 (1)
Dizziness (Nervous system disorders) | 51 (65) | 34 (40) | 0 (0)
Dysgeusia (Nervous system disorders) | 34 (41) | 27 (30) | 0 (0)
Headache (Nervous system disorders) | 102 (182) | 39 (47) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 11 (12) | 26 (37) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 18 (20) | 110 (132) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 90 (100) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 23 (24) | 12 (13) | 0 (0)
Insomnia (Psychiatric disorders) | 40 (45) | 27 (33) | 0 (0)
Dysuria (Renal and urinary disorders) | 23 (27) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 33 (46) | 11 (13) | 0 (0)
Proteinuria (Renal and urinary disorders) | 146 (293) | 13 (17) | 2 (2)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 32 (42) | 9 (11) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 64 (79) | 21 (24) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 64 (79) | 5 (15) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 (51) | 29 (32) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (30) | 17 (18) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 47 (49) | 220 (221) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 27 (32) | 8 (8) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 59 (79) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 49 (57) | 25 (34) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 77 (102) | 20 (23) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 (33) | 14 (14) | 0 (0)
Hypertension (Vascular disorders) | 288 (563) | 82 (107) | 2 (3)
Hypotension (Vascular disorders) | 28 (31) | 5 (5) | 1 (1)
White coat hypertension (Vascular disorders) | 1 (14) | 3 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03884101/Prot_SAP_000.pdf